CLINICAL TRIAL: NCT04253821
Title: Relationship Between the Tonus, Stiffness, and Elasticity of Head Posture Muscles and Pulmonary Capacity and Functional Capacity: a Myotonometric Assessment
Brief Title: Relationship Between Head Posture Muscles, Pulmonary Capacity and Functional Capacity: a Myotonometric Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cagtay Maden (Other)
Responsible Party: Sponsor-Investigator, Cagtay Maden, research assistant,physiotherapist, Hasan Kalyoncu University
Organization: Hasan Kalyoncu University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019/24
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Forward Head Posture; Muscle Tone; Muscle Stiffnes; Muscle Elasticty; Vital Capacity
Keywords: forward head posture; muscle elasticity
MeSH Terms: interventions — Muscle Tonus; Respiratory Physiological Phenomena

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forward head posture (Active Comparator)
  Interventions: Other: muscle tonus, stiffness and elasticity,six-minute walk test, Pulmonary function tests, The neck disability index
- Non-Forward head posture (Active Comparator)
  Interventions: Other: muscle tonus, stiffness and elasticity,six-minute walk test, Pulmonary function tests, The neck disability index

INTERVENTIONS:
Other: muscle tonus, stiffness and elasticity,six-minute walk test, Pulmonary function tests, The neck disability index — The muscle tonus, stiffness and elasticity of upper trapezius (UT), semispinalis capistis (SSC), pectoral muscles (PM) and sternocleidomastoideus muscles (SCM) were measured by using MyotonPro® device. Functional capacity was measured with six-minute walk test. Pulmonary function tests was evaluated with spirometer. The neck disability index (NDT) was applied. The forward head posture was determined by measurements of craniovertebral angle (CVA). Physical activity levels of participants were evaluated by Physical Activity Index (FIT).

SUMMARY:
Forward head posture (FHP) is known to have a large influence on respiratory function by weakening the respiratory muscles. This cross-sectional study is designed to examine the relationship between the tonus, stiffness, and elasticity of head posture muscles and pulmonary capacity. Sixteen FHP individuals and seventeen NFHP individuals were evaluated. The muscle tonus, stiffness and elasticity of upper trapezius (UT), semispinalis capistis (SSC), pectoral muscles (PM) and sternocleidomastoideus muscles (SCM) were measured by using MyotonPro® device. Functional capacity was measured with six-minute walk test. Pulmonary function tests was evaluated with spirometer. The neck disability index (NDT) was applied. The forward head posture was determined by measurements of craniovertebral angle (CVA). Physical activity levels of participants were evaluated by Physical Activity Index (FIT).

ELIGIBILITY:
Inclusion Criteria:

- the participants do not have any known pulmonary, systemic and muscular system disease and, any neurological symptoms and neck pain that affects daily living activities.

Exclusion Criteria:

* have headache and dizziness
* steroid use or muscle relaxants

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
muscle tonus, stiffness and elasticity | 1 day
  The measurements of muscle tone, stiffness and elasticity were made by using MyotonPro® device. Participants were seated on the chair and hands were placed on the knee, UT, SSC and SCM muscles were measured in this position. The pectoralis major muscle was measured in the supine position.
six-minute walk test. | 1 day
  Functional capacity was measured with six-minute walk test.
Vital Capacity | 1 day
  Pulmonary function tests was evaluated with spirometer.It is the volume of air in the lungs that varies between full inspiration and maximum expiration.
Forced Vital Capacity (FVC) | 1 day
  Pulmonary function tests was evaluated with spirometer.It is the volume of air that comes out with rapid and powerful exhalation following deep inspiratory. Healthy people can normally extract 80% of their lung volume in 6 seconds or less.
Forced Expiratory Volume in 1 Second (FEV1) | 1 day
  Pulmonary function tests was evaluated with spirometer.It is the volume of air released in the first second from the beginning of the difficult vital capacity maneuver. In general, it gives information about the restriction in major airlines. FEV1 / FVC ratio decrease shows obstruction, FEV1 shows the severity of obstruction.
Peak Expiratory Flow (PEF) | 1 day
  Pulmonary function tests was evaluated with spirometer.It is measured by the maximum exhalation maneuver following the maximum inspiration. It gives information about obstruction in large airways.
The neck disability index | 1 day
  The neck disability index was applied. the total score is 50. As the test score rises, disability increases.0-4 score no disability, 5-14 mild disability, 15-24 moderate degree, 25-34 severe disability, 35 and above completely disabled
Physical Activity Index | 1 day
  The FIT index was used to classify the individuals' physical activity levels. This research instrument used to classify and assign a score from 1 to 100 to a person's physical fitness level based on their frequency, intensity, and time engaged in physical fitness activities. The physical activity score was obtained by multiplying the frequency, intensity and time of the activity. According to the FIT score, the physical activity level is interpreted as 0-20 sedentary, 21-40 weak, 41-60 normal, 61-80 good and 81-100 very good.
Forward head posture assessment | 1 day
  Forward head posture was assessed by a goniometric method which is accepted as a reliable method. Participants were assessed in a relaxed sitting position. To measure the craniovertebral angle (CVA) of FHP, the center of the goniometer is placed at the level of the orifice of the external ear with the fixed arm pointing vertically towards the ceiling and the moving arm against the subject's 7th neck bonee.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu Universty, Gaziantep, Şahinbey, Turkey (Türkiye)